CLINICAL TRIAL: NCT05958667
Title: Randomized Controlled Trial to Assess Innovative Smoking Cessation Services for Young Adults in Texas
Brief Title: Quitxt Mobile Text Messaging Cessation Research Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other); The University of Texas at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC20230473H
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation
Keywords: Quitxt; Young adults; Latinos
MeSH Terms: conditions — Smoking Cessation | interventions — Choline O-Acetyltransferase

STUDY DESIGN:
Intervention Model Description: A two-group parallel randomized controlled trial with 1,200 Spanish- and English-speaking young Latino adult smokers in South Texas (ages 18-29) to assess the effects of Quitxt on smoking cessation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quitxt bilingual text messaging and chat (Experimental): Culturally and linguistically tailored, bilingual text messaging or chat mobile app.
  Our text messaging or chat intervention will include messaging options in which users can text or message a code when they are craving a cigarette or at risk of relapse and immediately receive text or social media messages to help them avoid smoking. The social media content also will include opportunities for users to repeatedly visit key content pages and receive immediate support when experiencing cravings, stress, bad mood, or when feeling at risk of smoking.
  Interventions: Behavioral: Quitxt text messaging or Chat
- Usual care (Other): Abbreviated text messaging with smoking cessation-related content and referral to the Texas Department of State Health Services (TDSHS) cessation program Yes Quit (www.yesquit.org) available to smokers seeking help quitting. The abbreviated text messaging will include general information on smoking harms and benefits of cessation, and baseline data collection and follow-up assessments.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Quitxt text messaging or Chat — Mobile intervention using proven social cognitive, motivational interviewing, and brief intervention methods for promoting behavior change - blends bilingual text and social media messaging for smoking cessation tailored to the language and culture of young adult smokers in our vulnerable region of South Texas.
  Other Names: Culturally appropriate mobile smoking cessation proram
  Arms: Quitxt bilingual text messaging and chat
Other: Usual care — Abbreviated text messaging with smoking cessation-related content and referral to the Texas Department of State Health Services (TDSHS) cessation program Yes Quit.
  Other Names: Abbreviated text messaging with smoking cessation-related content
  Arms: Usual care

SUMMARY:
The health benefits of smoking cessation by age 30 are much greater than cessation later in life, including gaining 10 years of life, compared with those who continue to smoke. The goal of the proposed study is to evaluate the effectiveness of the bilingual and culturally tailored Quitxt mobile cessation intervention. Quitxt provides interactive messages through texts or chat with visual and video content employing theory- and evidence-based techniques to prompt and sustain cessation. The study will recruit 1,200 Latino young adult smokers aged 18-29 who enroll and agree to make quit attempts, with half randomly assigned (like flipping a coin) to receive Quitxt and half to abbreviated text messages with smoking cessation-related content and referral to the Texas Department of State Health Services cessation program Yes Quit (which has diverse formats, but not explicitly tailored for young Latino adults in South Texas). Participants respond to baseline and follow-up assessments at one, three and six months after their enrollment, and those who report cessation will be asked to provide saliva samples to confirm they quit smoking. The sample size will be sufficient to detect expected higher cessation rates in those who are enrolled in Quitxt than those who are enrolled in Texas DSHS Yes Quit. The investigators will publish results in scientific journals, report them at scientific and community meetings, share them on social media, and publicize them widely. This study has the potential to advance public health by evaluating the effectiveness of a scalable, easily disseminated and adaptable intervention to help young adults, especially Latinos, quit smoking and reduce smoking-related cancer and chronic disease morbidity and mortality and their associated healthcare costs.

DETAILED DESCRIPTION:
Despite major advances in tobacco control and treatment, tobacco use remains the single largest preventable cause of morbidity and mortality in the US. Smoking prevalence is highest among Texas young adults (ages 18-29) and even higher among those with less than a high-school education and those living in rural areas and at or below the poverty level, such as Latinos. About 19.2% of Latinos ages 18-29 in the study areas are current smokers placing them at higher risk of cancer and other tobacco-related morbidity and mortality. Young adults are heavy users of smartphones, text messaging, social media chats and other mobile social media, providing a remarkable opportunity for innovation in the delivery of health promotion services to reduce health disparities in this large and rapidly growing racial/ethnic population. New social media have an extraordinary theoretical potential for assisting smoking cessation by providing peer modeling and eliciting social reinforcement for behavior change. The goal of this project is to experimentally evaluate Quitxt, a culturally appropriate mobile smoking cessation program. Quitxt - launched by an interdisciplinary research team using proven social cognitive, motivational interviewing, and brief intervention methods for promoting behavior change - blends bilingual text and social media messaging for smoking cessation tailored to the language and culture of young adult smokers in the vulnerable region of South Texas. Quitxt has not been tested in a research study, as its creation as an evidence-based cancer prevention service for young adult smokers was supported by the Cancer Prevention and Research Institute of Texas (CPRIT). To study the effects of Quitxt, the study team will recruit 1,200 young adult (ages 18-29) Latino Spanish- and English-speaking smokers over the 5-year study interval in South Texas. A two-group parallel randomized controlled trial will be conducted to compare rates of smoking cessation: 1) the intervention group will receive the innovative Quitxt text messaging or the chat mobile service; and 2) the usual care group will receive abbreviated text messaging with smoking cessation-related content and referral to the Texas Department of State Health Services (TDSHS) cessation program Yes Quit (www.yesquit.org). The investigators will measure effects online at time of enrollment and again at one, three and six months later. The investigators will validate reports of smoking cessation via biological tests, for those who report smoking cessation at one, three and six-month follow-ups. The investigators hypothesize that the group receiving the Quitxt intervention will achieve significantly higher smoking cessation rates than the group receiving usual care. This study will expand research on the health of young adult Latinos by testing an innovative, mobile, culturally, and linguistically appropriate intervention to reduce smoking among young adult Latino smokers by enhancing their skills development, competence, and self-efficacy to initiate and maintain cessation. Moreover, this study will advance public health by testing the effectiveness of a scalable, evidence-based, easily disseminated, and adaptable intervention with potentially broad national reach to help young adults stop smoking and reduce smoking-related cancer and chronic disease morbidity and mortality and their associated healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. Latinos
2. aged 18-29 years;
3. smoking at least one cigarette/day ≥3 days/week;
4. interested in quitting;
5. willing to provide follow-up data;
6. are not simultaneously participating in a cessation program;
7. own a cell phone or smartphone;
8. are able to send and receive text messages and access the Internet;
9. reside in the study area; and
10. able to provide informed consent to participate in the study.

Exclusion Criteria:

1. are not interested in quitting;
2. are unable to provide consent due to a mental, emotional, or physical handicap that keep them from understanding the consent information;
3. do not own a cell phone with text and Internet capabilities;
4. are unable to respond to text messages and questions or unable to view the study mobile webpages/YouTube videos (i.e., if they are blind, deaf); or
5. are planning to move from the study area within the study time span.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation | 6 months
  Measure of smoking cessation (7-day point prevalence abstinence)self-reported and biochemically verified.

SECONDARY OUTCOMES:
Smoking cessation assessment | 1 month and 3 months
  Measure of smoking cessation (7-day point prevalence abstinence)self-reported and biochemically verified.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Chalela, DrPH, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Annual presentation at a national conference is expected. Community Presentations/Forums for young adult organizations and groups, public health and clinical practitioners, and the community at large.
  Educational presentations and infographics about the importance of quitting smoking aimed at colleges, technical schools, community stakeholders, at health fairs or at in-person and/or virtual educational sessions organized with the study team's community partners.
  Submission to scientific journals Communications, American Journal of Health Promotion, Tobacco Control, and other scientific periodicals to disseminate findings including Quitxt text messaging and chat development and implementation and report experimental results based on follow-up assessments.
  Via the Institute for Health Promotion Research home website; its institutional e-newsletters; and its Salud America! (SA!) national network.
Supporting Information: Study Protocol, SAP
Time Frame: At study completion when summary data are published or otherwise made available
Access Criteria: Institute for Health Promotion Research home website; its institutional e-newsletters; and its Salud America! (SA!) national network.
URL: http://ihpr.uthscsa.edu